CLINICAL TRIAL: NCT05762367
Title: MR Lymphatic Imaging in Idiopathic Intracranial Hypertension
Brief Title: MR Lymphatic Imaging in Idiopathic Intracranial Hypertention
Acronym: LYMPHIMAGIIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: C22-13; 2022-A01422-41 (Other: IDRCB)
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: Dural venous stenoses; MRI; Vessel Wall Imaging; Headache; Papilledema
MeSH Terms: conditions — Pseudotumor Cerebri; Headache; Papilledema

STUDY DESIGN:
Intervention Model Description: 20 patients with IIH and 20 volunteers paired on age (20-40 yo) and gender will be prospectively enrolled in the study
Who Masked: Investigator, Outcomes Assessor
Masking Description: MRI will be pseudo-anonymised and blindly analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with IIH (Experimental): Female patients with IIH between 20 and 40 years old
  Interventions: Diagnostic Test: 3T MRI with Gadobutrol injection
- Healthy volunteers (Active Comparator): Female healthy volunteers between 20 and 40 years old
  Interventions: Diagnostic Test: 3T MRI with Gadobutrol injection

INTERVENTIONS:
Diagnostic Test: 3T MRI with Gadobutrol injection — MRI will be performed in all participants before and after Gadobutrol injection

SUMMARY:
In the brain and its borders, blood vessels coexist with lymphatic vessels exclusively in the dura mater, the outermost layer of meninges. Dural lymphatics are present in various vertebrate species, including humans, and a cluster of experimental studies in the mouse strongly suggest their relevance in the pathophysiology of chronic and acute neurological disorders in humans. Demonstrating this assumption is however still at stake and the lymphatic regulatory mechanisms involved remain poorly characterized.

Our main objective is to assess dural lymphatics contribution to the pathophysiology of a rare neurological disorder: idiopathic intracranial hypertension (IIH). In IIH patients, intracranial hypertension causes severe headache and visual loss and is associated with a stenosis of dural sinuses and abnormal retention of fluids in the central nervous system. Angioplasty treatment by stent placement into venous sinuses is frequently followed by recurrent stenosis suggesting that, in addition to the blood vessels, the duro-lymphatic environment contributes to disease progression.

Several studies have found hot spots of lymphatic uptake at confluence points between cerebral veins and dural sinuses. Based on this premise, the investigators predict a causal link between lymphatic and venous behavior around dural sinuses and the remodeling of dural lymphatics in neurovascular conditions such as IIH.

Our approach will combine radiological observations from human patients with experimental analyses in mouse models.

The investigators have recently developed a technique of high resolution vessel wall imaging to explore and compare the lymphatic networks between individuals. This advanced MR-imaging technique has been validated through a translational study comparing the lymphatic networks in mice and humans (Jacob et al. 2022, JExpMed). Using this tool, the investigators aim to monitor dural lymphatic and sinus wall abnormalities in patients with IIH. In this view, cohorts of IIH patients and controls without neurological disorders (n = 20/cohort) will be scanned by MRI to perform high resolution vessel wall imaging of the dural lymphatics, sinus and cerebral veins.

DETAILED DESCRIPTION:
Fluid retention in idiopathic intracranial hypertension (IIH) (Lenck, Neurology 2018) preferentially occur at the "hot spots" of the dural lymphatic system described in mice (Ahn, Nature 2019; Ma, Nat Commun 2017; Louveau, Nat Neurosci. 2018). While the pathophysiological mechanisms of IIH are still unknown, dural venous stenoses are constant and endovascular treatment by stenting allow to decrease the intracranial pressure in most cases, suggesting a crucial role of these stenoses in the pathological process of IIH. However, the cause of dural venous sinsu stenoses are still unknown. IIH corresponds to a paradigmatic model of neurological disorder associating vascular and fluid dysfunction, since raised intracranial pressure and stenosis of the dural venous sinuses are in constant association. Dural venous stenoses are located at the transverse sinus-sigmoid sinus junction, a lymphatic reuptake point or 'hot spot', in mice. The pathological process leading to the progressive obstruction of the vein seems to directly affect the wall of the dural sinus and only secondarily its lumen (Lenck, Neurology 2018; Lenck, AJNR 2021; Lenck, Neurosurgery 2017; Kedra, JNNP 2021). Impaired lymphatic reuptake could also contribute to this pathology as suggested by the accumulation of fluid at the level of the cribriform plate, or at the Meckel's cave. Thus, the association between cerebral venous outflow obstruction and CSF accumulation in the dura mater at the hotspots of the lymphatic system suggests impaired dural lymphatic system and veno-lymphatic relationships in IIH.

Since 2017, and the first demonstration by MRI of the dural lymphatics in humans by Absinta (Absinta, Elife. 2017), VWI (Vessel Wall Imaging) techniques have been significantly improved in terms of resolution allowing an analysis of the cerebral vessel wall (Xie et al. Magn Reson Med. 2016). These techniques were mainly developed in the context of arterial wall abnormalities but have never been applied to the study of the dural venous wall and its lymphatics. The 3D T1 SPACE (variable flip angle turbo spin echo) - DANTE (delay alternating with nutation for tailored excitation) sequence has been recently developed and allows to improve the suppression of the intravascular signal and consequently to improve the resolution of the vessel wall imaging (Xie et al. Magn Reson Med. 2016). In collaboration with Siemens, our team has further developed and improved this advanced VWI technique and performed a translational comparative study comparing the dural lymphatic network between humans and mice to validate its preliminary results (Jacob, J. Exp. Med 2022). This study allowed to characterize the entire dural lymphatic network with high resolution and in three dimensions, as well as its connections with the cervical lymph nodes in humans. Furthermore, the investigators firstly demonstrated the presence of a ventral lymphatic network around the cavernous sinus. Our results seem superior to previous radiological protocols for qualitative and large field analysis of the parasinus and its lymphatics. Image processing by dedicated segmentation software (3D-Slicer) allows a three-dimensional reconstruction of the veno-lymphatic network in humans but also its quantitative analysis. This represents a major scientific breakthrough allowing objective comparisons of these networks between pathologies.

IIH is a still mysterious and poorly known entity at the frontiers of neurology, neurosurgery and ophthalmology. It affects young women of childbearing age and can lead to a major deterioration in the quality of life through headaches, visual impairment or even the blindness that it can cause. All available treatments (Acetazolamide, CSF diversion, venous stent) are active on the symptoms of the disease but do not target its cause. Their effectiveness is limited, they are invasive and associated with significant risks and adverse effects. More effective and less invasive therapies, directly targeting the biological cause of IIH, therefore represent a major medical challenge.

However, a prerequisite before considering such approach is to understand the pathophysiological bases underlying IIH. Our project combines innovative experimental approaches in surgery and imaging on murine models with the previously described development of lymphatic imaging in humans in patients with IIH and controls. The ultimate goal of our research is to open therapeutic avenues with realistic potential to improve the prognosis of patients with IIH.

In this study the investigators will enroll 20 female patients with IIH and 20 female healthy volunteers between 20 and 40 years old.

Our primary objective is to compare the anatomy of the dural lymphatic network in patients with IIH compared to healthy subjects.

Our secondary objectives are:

* Characterization in high resolution VWI imaging of dural venous sinus stenoses in IIH
* Morphometric study of the cervical lymphatic network in patients with IIH compared to healthy subjects.
* Comparison of the volume of the different compartments of the skull between patients with IIH and healthy volunteers (cerebral volume, intraventricular CSF volume (lateral ventricles), intradural venous volume)

ELIGIBILITY:
Inclusion Criteria:

* For all participants:

Age > 18 years and ≤ 40 years female gender Absence of previous neurosurgical or endovascular neurological history Participant able to express her consent Medical insurance

* For participants with IIH No required criterion of severity or evolution of IIH Definite diagnosis of IIH according to Dandy's modified criteria. All of the following criteria must be met and verified by medical reports or certificates from a neurologist, especially the value of the CSF opening pressure measured during the lumbar puncture must be clearly noted on the reports

  * History of papilledema
  * Normal neurological examination, except for paralysis of the VIth cranial nerve
  * Neuroimaging: normal cerebral parenchyma without hydrocephalus, intracranial expansive process, or structural anomaly, and absence of meningeal contrast enhancement in MRI without and with contrast product. A venous angio-MRI is necessary in atypical patients; if MRI is unavailable or contraindicated, a brain scan without and with contrast product can be done in combination with a venous angioscan with contrast injection
  * Normal CSF composition
  * High CSF opening pressure (≥ 25 cm of water) obtained from a lumbar puncture performed in lateral decubitus
* For healthy volunteers No previous history of neurological or neurosurgical disorder

Exclusion Criteria:

* For all participants Pregnant or breastfeeding woman Contraindication to cerebral MRI: metallic implant, pacemaker, artificial heart valve, cerebral vascular malformation, aneurysm clips, metallic fragments, artificial implants, peripheral or neural pacemaker, insulin pump, intravenous catheter, epilepsy , metallic contraceptive device, claustrophobia, refusal to be informed in case of abnormal MRI (with a significant medical abnormality) Hypersensitivity to the active substance of the contrast agent or to any of the excipients (Sodium calcobutrol, Trometamol, 1N hydrochloric acid (pH adjustment), Water for injections) lumbar puncture in the month preceding the brain MRI Neurological tumoral, degenerative, vascular, inflammatory or progressive pathology Renal or hepatic impairment MRI with gadolinium injection performed in the 7 days preceding the inclusion visit Person subject to a measure of legal protection (safeguard of justice, curatorship, guardianship), deprived of liberty by judicial or administrative decision
* For participants with IIH Participants with a probable but not definite diagnosis of IIH according to the Dandy modified criteria
* For healthy volunteers Chronic headaches (>15 days per month) Uncorrected and/or unlabeled visual symptoms (visual blurriness, diplopia, visual eclipses, papilledema, optic atrophy)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-05-11 (Actual)

PRIMARY OUTCOMES:
Morphometric study of the dural lymphatic network in patients with IIH vs controls | Immediate
  Measurement of the dural lymphatic network volume (mm3) in patients with IIH vs controls

SECONDARY OUTCOMES:
Characterization of lateral sinus stenoses using high resolution vessel wall imaging in patients with IIH | Immediate
  Measurement of the volume of the dural lymphatic vessels at the transverse-sigmoid junction in patients with IIH vs control Measurement of the thickness of the parasinus at the transverse-sigmoid junction in patients with IIH vs control Measurement of the stenosis (ratio intraluminal diameter at the level of the stenosis and intraluminal diameter of the transverse sinus upstream) in patients with IIH Presence of intraluminal granulation in patients with IIH vs control Qualitative analysis of dural venous stenoses in patients with IIH
Morphometric study of the cervical lymphatic network in patients with IIH vs controls | Immediate
  Comparison of the volume of the cervical lymph nodes in patients with IIH vs controls
Comparison of the volumes of the different compartments of the skull in patients with IIH vs controls | Immediate
  Brain volume in patients with IIH vs controls Intraventricular CSF volume of the lateral ventricles in patients with IIH vs controls Intradural venous volume in patients with IIH vs controls

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neuroradiologie, Groupe Hospitalier Pitié Salpêtrière, Paris, France, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn JH, Cho H, Kim JH, Kim SH, Ham JS, Park I, Suh SH, Hong SP, Song JH, Hong YK, Jeong Y, Park SH, Koh GY. Meningeal lymphatic vessels at the skull base drain cerebrospinal fluid. Nature. 2019 Aug;572(7767):62-66. doi: 10.1038/s41586-019-1419-5. Epub 2019 Jul 24. PMID 31341278
- [Background] Lenck S, Radovanovic I, Nicholson P, Hodaie M, Krings T, Mendes-Pereira V. Idiopathic intracranial hypertension: The veno glymphatic connections. Neurology. 2018 Sep 11;91(11):515-522. doi: 10.1212/WNL.0000000000006166. PMID 30201744
- [Background] Ma Q, Ineichen BV, Detmar M, Proulx ST. Outflow of cerebrospinal fluid is predominantly through lymphatic vessels and is reduced in aged mice. Nat Commun. 2017 Nov 10;8(1):1434. doi: 10.1038/s41467-017-01484-6. PMID 29127332
- [Background] Louveau A, Herz J, Alme MN, Salvador AF, Dong MQ, Viar KE, Herod SG, Knopp J, Setliff JC, Lupi AL, Da Mesquita S, Frost EL, Gaultier A, Harris TH, Cao R, Hu S, Lukens JR, Smirnov I, Overall CC, Oliver G, Kipnis J. CNS lymphatic drainage and neuroinflammation are regulated by meningeal lymphatic vasculature. Nat Neurosci. 2018 Oct;21(10):1380-1391. doi: 10.1038/s41593-018-0227-9. Epub 2018 Sep 17. PMID 30224810
- [Background] Lenck S, Nicholson P. Cerebral Venous Wall Diseases: The Other Side of the Picture. AJNR Am J Neuroradiol. 2021 Jan;42(2):297-298. doi: 10.3174/ajnr.A6914. Epub 2021 Jan 7. No abstract available. PMID 33414232
- [Background] Lenck S, Vallee F, Labeyrie MA, Touitou V, Saint-Maurice JP, Guillonnet A, Tantot A, Crassard I, Bernat AL, Houdart E. Stenting of the Lateral Sinus in Idiopathic Intracranial Hypertension According to the Type of Stenosis. Neurosurgery. 2017 Mar 1;80(3):393-400. doi: 10.1227/NEU.0000000000001261. PMID 27218234
- [Background] Kedra A, Lahlouh M, Shotar E, Chenoune Y, Boistard L, Boussac A, Shor N, Savatovsky J, Hage R, Touitou V, Nicholson P, Clarencon F, Piotin M, Blanc R, Lenck S. Global collapse of the dural sinuses after venous stenting in idiopathic intracranial hypertension. J Neurol Neurosurg Psychiatry. 2021 Dec;92(12):1363-1364. doi: 10.1136/jnnp-2020-325717. Epub 2021 Jun 24. No abstract available. PMID 34168084
- [Background] Absinta M, Ha SK, Nair G, Sati P, Luciano NJ, Palisoc M, Louveau A, Zaghloul KA, Pittaluga S, Kipnis J, Reich DS. Human and nonhuman primate meninges harbor lymphatic vessels that can be visualized noninvasively by MRI. Elife. 2017 Oct 3;6:e29738. doi: 10.7554/eLife.29738. PMID 28971799
- [Background] Xie Y, Yang Q, Xie G, Pang J, Fan Z, Li D. Improved black-blood imaging using DANTE-SPACE for simultaneous carotid and intracranial vessel wall evaluation. Magn Reson Med. 2016 Jun;75(6):2286-94. doi: 10.1002/mrm.25785. Epub 2015 Jul 8. PMID 26152900
- [Background] Jacob L, de Brito Neto J, Lenck S, Corcy C, Benbelkacem F, Geraldo LH, Xu Y, Thomas JM, El Kamouh MR, Spajer M, Potier MC, Haik S, Kalamarides M, Stankoff B, Lehericy S, Eichmann A, Thomas JL. Conserved meningeal lymphatic drainage circuits in mice and humans. J Exp Med. 2022 Aug 1;219(8):e20220035. doi: 10.1084/jem.20220035. Epub 2022 Jul 1. PMID 35776089